CLINICAL TRIAL: NCT06233552
Title: Smart Digital Denture Conversion (SDDC), a Technique for Full Arch Immediate Loading: A Randomized Trial
Brief Title: Smart Digital Denture Conversion (SDDC), a Technique for Full Arch Immediate Loading
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, yasmine Elsherbeeny, lecturer at the prosthodontics department, faculty of dentisrty, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: FDASU-Rec IR 102305
Record Dates: First submitted 2023-12-18; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Complete Edentulism
Keywords: immediate loading; denture conversion; full arch implant rehabilitation

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- conventional denture conversion (Active Comparator): a conventional denture conversion will be done following the conventional fabrication technique.
  Interventions: Procedure: conventional denture conversion
- digital denture conversion (Experimental): An alternative workflow for construction of the fixed interim requires impressions, model production, and jaw relation records then digitizing all these data then designing and milling the restoration.
  Interventions: Procedure: digital denture conversion

INTERVENTIONS:
Procedure: conventional denture conversion — conventional workflow usually done to do immediate loading for full arch implant cases
  Arms: conventional denture conversion
Procedure: digital denture conversion — An alternative workflow for construction of the fixed interim requires impressions, model production, and jaw relation records then digitizing all these data then designing and milling the restoration.
  Arms: digital denture conversion

SUMMARY:
This study presents a smart digital approach to design and construct a screw retained immediately loaded full arch implant supported bridge based on the pre-treatment complete denture.

DETAILED DESCRIPTION:
After intra oral scanning of the ridge form, implant positions, the denture is used to scan the intermaxillary relation and tooth positions and the fixed interim is designed and milled from PMMA. This technique is applicable when a single arch is treated or for bimaxillary implant rehabilitation cases. In this study 30 patients were grouped into two groups; group I in which a converted denture was made conventionally and Group II in which a converted denture was made digitally. General satisfaction, chair side working time, and esthetic outcome of the prostheses were recorded and quantified with a verbal rating scale following insertion of implant-supported prosthesis.

ELIGIBILITY:
Inclusion Criteria:

* -Nonsmokers
* Free from any systemic disease
* Non-bruxers
* With sufficient quality and quantity of bone
* Prepared to comply with the follow-up and maintenance program

Exclusion Criteria:

* - Patients with bad oral hygiene.
* Patients with limited mouth opening.
* Vulnerable groups.
* Uncooperative patients.

Ages: 50 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2023-03-01 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Patient general satisfaction questionnaire | through study completion within 6 months
  General satisfaction with a verbal rating scale range from 0 to 5, as 0 denotes the lowest value (worst) and 5 the highest value (best), following insertion of implant-supported prosthesis.

SECONDARY OUTCOMES:
chair side working time questionnaire | through study completion within 6 months
  the procedure working time with a verbal rating scale range from 0 to 5, as 0 denotes the lowest value (worst) and 5 the highest value (best), following insertion of implant-supported prosthesis.
esthetic satisfaction questionnaire | through study completion within 6 months
  esthetic outcome of the prostheses with a verbal rating scale range from 0 to 5, as 0 denotes the lowest value (worst) and 5 the highest value (best), following insertion of implant-supported prosthesis.

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

DOCUMENTS (2):
  • Study Protocol (2023-11-01): https://cdn.clinicaltrials.gov/large-docs/52/NCT06233552/Prot_000.pdf
  • Statistical Analysis Plan (2023-10-27): https://cdn.clinicaltrials.gov/large-docs/52/NCT06233552/SAP_001.pdf